CLINICAL TRIAL: NCT01941940
Title: A National, Open-Label, Single-Arm, Phase IIIb Study to Evaluate the Efficacy of Weekly Tocilizumab Subcutaneous, Administered as Monotherapy or in Combination With Methotrexate and/or Other DMARDs in Rheumatoid Arthritis (RA) Patients
Brief Title: A Study to Evaluate Efficacy of Tocilizumab Administered as Monotherapy or in Combination With Methotrexate and/or Other Disease Modifying Antirheumatic Drugs (DMARDs) in Rheumatoid Arthritis (RA) Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28699; 2013-001569-17 (EudraCT Number)
Record Dates: First submitted 2013-09-02; First posted 2013-09-13 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Antirheumatic Agents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tocilizumab (Experimental): Tocilizumab at a fixed dose of 162 milligrams (mg) will be administered as subcutaneous (SC) injection alone or along with methotrexate and/or other non-biological DMARDs irrespective of body weight, once every week for a total of 52 weeks. After 52-weeks of treatment, at the discretion of the treating physician, participants can continue the study treatment with SC tocilizumab until it becomes commercially available in Italy.
  Interventions: Drug: Tocilizumab; Drug: DMARDs

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab at a fixed dose of 162 mg as SC injection will be administered once every week.
  Other Names: RoActemra
Drug: DMARDs — Non-biologic DMARDs according to standard of care, at a stable dose that was initiated at least 4 weeks prior to baseline.

SUMMARY:
This open-label, single arm, Phase 3b study will evaluate the efficacy of tocilizumab (RoActemra), administered as monotherapy or in combination with methotrexate and/or other DMARDs, in participants with moderate to severe active RA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active RA according to the revised (1987) ACR criteria or EULAR/ACR (2010) criteria
* Moderate to severe RA (CDAI at least [>/=] 10 and DAS28 >/=3.2) at screening
* Tumor necrosis factor inhibitors-inadequate responder (TNF-IR), methotrexate-inadequate responder (MTX-IR), and/or DMARDs-inadequate responder (DMARDs-IR)
* Oral corticosteroids (less than or equal to [</=] 10 mg per day prednisone or equivalent) and non-steroidal anti-inflammatory drugs (NSAIDs; up to the maximum recommended dose) are permitted if on a stable dose regimen for >/=4 weeks prior to baseline
* Permitted non-biologic DMARDs are allowed if at a stable dose for >/=4 weeks prior to baseline
* Receiving treatment on an outpatient basis, not including tocilizumab
* Females of childbearing potential and males with female partners of childbearing potential must agree to use a reliable means of contraception for at least 3 months following the last dose of tocilizumab

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 12 months following baseline
* Rheumatic autoimmune disease other than RA; secondary Sjögren's syndrome with RA is permitted
* Functional Class IV as defined by the ACR Classification of Functional Status in RA
* Diagnosis of juvenile idiopathic arthritis or juvenile RA and/or RA before the age of 16
* Prior history of or current inflammatory joint disease other than RA
* Exposure to tocilizumab (either intravenous [IV] or SC) at any time prior to baseline
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening
* Previous treatment with any cell-depleting therapies
* Intra-articular or parenteral corticosteroids within 4 weeks prior to baseline
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine (including uncontrolled diabetes mellitus), or gastrointestinal disease
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks of screening
* Active tuberculosis (TB) requiring treatment within the previous 3 years
* Positive for hepatitis B surface antigen or hepatitis C antibody
* Primary or secondary immunodeficiency (history of or currently active)
* Evidence of active malignant disease, malignancies diagnosed within the previous 10 years (except for basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured), or breast cancer diagnosed within the previous 20 years
* Pregnant or breast feeding women
* Neuropathies or other conditions that might interfere with pain evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2015-09-09 (Actual); Study Completion 2016-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (49):
- Italy (49):
  - Uni Degli Studi Di L Aquila; Cattedra Di Reumatologia - Dept. Di Medicina Interna E San, Coppito, Abruzzo
  - P. O. Spirito Santo - Asl Pescara; U.O. Complessa Di Reumatologia, Pescara, Abruzzo
  - Ospedale Regionale Umberto Parini; Reparto Endocrinologia e Diabetologia - Amb. Reumatologia, Aosta, Aosta Valley
  - Azienda Ospedaliera Policlinico; Servizio Reumatologia, Bari, Apulia
  - ASL Lecce- Presidio Ospedaliero di Casarano-Servizio di Reumatologia ed Osteoporosi, Casarano (LE), Apulia
  - Ospedali Riuniti di Foggia; Dipartimento Medicina Interna Reumatologia, Foggia, Apulia
  - Ospedali Riuniti Di Foggia; Struttura Di Reumatologia, Foggia, Apulia
  - Azienda Ospedaliera Bianchi Melacrino Morelli; Unità Operativa di Reumatologia, Reggio Calabria, Calabria
  - Az. Ospedaliera S. Giuseppe Moscati; Dip. Med. Gen. Struttura Semplice Reumatologia, Avellino, Campania
  - Azienda Ospedaliera Rummo; Divisione Di Reumatologia, Benevento, Campania
  - Azienda Ospedaliera A. Cardarelli; Medicina III - Divisione di Reumatologia, Napoli, Campania
  - Policlinico Universitario-II Università di Napoli; Reumatologia, Napoli, Campania
  - Osp Riuniti S.Giovanni di Dio e Ruggi d'Aragona; Rep. Medicina Interna, Salerno, Campania
  - Irccs Fondazione Salvatore Maugeri-Istituto Scientifico Di Telese;U.O. Riabilitazione Reumatologica, Telese Terme, Campania
  - A.O.U Policlinico S. Orsola Malpighi di Bologna U.O di Medicina Interna Borghi - Pad.2, Bologna, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Reumatologia, Modena, Emilia-Romagna
  - Arcispedale Santa Maria Nuova; Reumatologia, Reggio Emilia, Emilia-Romagna
  - Policlinico Univ. Uni Degli Sudi Di Udine; Clinica Di Reumatologia, Udine, Friuli Venezia Giulia
  - Policlinico Campus Bio-Medico Di Trigoria; Medicina Clinica E Reumatologia, Rome, Lazio
  - Policlinico Tor Vergata; Divisione Di Reumatologia, Rome, Lazio
  - Ospedale S.Pietro Fatebenefratelli; Divisione di Reumatologia, Rome, Lazio
  - Ospedale La Colletta; Reparto Di Reumatologia, Arenzano, Liguria
  - Università Degli Studi Di Genova - Dimi; Reumatologia, Genoa, Liguria
  - Ospedale San Paolo; Divisione di Reumatologia, Savona, Liguria
  - Asst Papa Giovanni XXIII; Dh Reumatologia, Bergamo, Lombardy
  - Ospedale Civile "La Memoria" Di Gavardo;Immunoematologia Trasfusionale-Allergologia E Reumatologia, Gavardo, Lombardy
  - Ospedale Di Magenta Fornaroli; U.O. Di Reumatologia, Magenta, Lombardy
  - Asst Centro Specialistico Ortopedico Traumato-Logico Gaetano Pini/Cto; Divisione Di Reumatologia, Milan, Lombardy
  - Ospedale Maggiore Policlinico; Unità Operativa Complessa di Allergologia e Immunologia Clinica, Milan, Lombardy
  - ASST FATEBENEFRATELLI SACCO; Reumatologia (Sacco), Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Reumatologia, Milan, Lombardy
  - ASST DI MONZA; Reumatologia (Medicina I), Monza, Lombardy
  - Irccs Policlinico San Matteo; Reumatologia Adulti, Pavia, Lombardy
  - ASST DI VIMERCATE; Medicina Generale, Vimercate, Lombardy
  - Azienda Ospedaliera Maggiore Della Carita; Day Hospital Immunologia, Novara, Piedmont
  - Azienda Ospedaliera San Giovanni Battista; Reparto Reumatologia, Turin, Piedmont
  - Ordine Mauriziano Ospedale Umberto I; Centro Di Reumatologia, Turin, Piedmont
  - A.O. Universitaria Policlinico Monserrato Di Cagliari; Reumatologia I, Cagliari, Sardinia
  - Azienda Ospedaliero Universitaria di Sassari; UOC Reumatologia, Sassari, Sardinia
  - Ospedale Vittorio Emanuele Ii; U.O. Reumatologia Clinica Medica Condorelli, Catania, Sicily
  - Azienda Osped. Univ. Policlinico G. Martino; Centro Prevenzione E Cura Osteoporosi, Messina, Sicily
  - Arnas Ospedale Civico; Medicina Interna II, Palermo, Sicily
  - Ospedale Regionale Torrette; SOD Clinica Medica del Dipartimento di Medicina Interna e Specialisti, Ancona, The Marches
  - Ospedale Murri - Universita Politecnica Delle Marche; Clinica Reumatologica Ii, Iesi, The Marches
  - Ospedale Careggi Villa Monnatessa ; Sezione Di Reumatologia, Florence, Tuscany
  - Az. Osp. Pisana Ospedale S. Chiara; U.O. Di Reumatologia, Pisa, Tuscany
  - Osp S. Maria Misericordia Dip. Medicina Clinica Sperimentale Cattedra Reumatologia, Perugia, Umbria
  - Azienda Ospedaliera Universitaria Borgo Trento; Dipartimento di Medicina Sezione di Reumatologia, Verona, Veneto
  - Policlinico G.B. Rossi; Divisione Immunologia Clinica Sperimentale Medicina B, Verona, Veneto

REFERENCES:
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Devenport J, Petho-Schramm A. Effects of concomitant glucocorticoids in TOZURA, a common-framework study programme of subcutaneous tocilizumab in rheumatoid arthritis. Rheumatology (Oxford). 2019 Jun 1;58(6):1056-1064. doi: 10.1093/rheumatology/key393. PMID 30649524
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Bernasconi C, Petho-Schramm A. Subcutaneous tocilizumab in rheumatoid arthritis: findings from the common-framework phase 4 study programme TOZURA conducted in 22 countries. Rheumatology (Oxford). 2018 Mar 1;57(3):499-507. doi: 10.1093/rheumatology/kex443. PMID 29244149

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of a total of 288 participants screened, 60 participants were excluded due to screening failure and 1 participant did not receive study treatment based on investigator's decision. Thus, total 227 participants were included in the study.
Groups:
- Tocilizumab: Tocilizumab at a fixed dose of 162 milligrams (mg) was administered as subcutaneous (SC) injection alone or along with methotrexate and/or other non-biological Disease-Modifying Antirheumatic Drugs (DMARDs) irrespective of body weight, once every week for a total of 52 weeks. After 52-weeks of treatment, at the discretion of the treating physician, participants could continue the study treatment with SC tocilizumab until it became commercially available in Italy (maximum up to 638 days).
Period: Overall Study
Arm/Group | Tocilizumab
Started | 227
Completed | 194
Not Completed | 33
Not completed — Adverse Event | 11
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 15
Not completed — Death | 1
Not completed — Other | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all recruited participants who received at least one dose of SC tocilizumab.
Groups:
- Tocilizumab: Tocilizumab at a fixed dose of 162 mg was administered as SC injection alone or along with methotrexate and/or other non-biological DMARDs irrespective of body weight, once every week for a total of 52 weeks. After 52-weeks of treatment, at the discretion of the treating physician, participants could continue the study treatment with SC tocilizumab until it became commercially available in Italy (maximum up to 638 days).
Arm/Group | Tocilizumab
Number analyzed (Participants) | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 24
Description: The CDAI is a numerical sum of 4 outcome parameters: tender joint count (TJC) and swollen joint count (SJC) based on a 28-joint assessment, patient's global assessment of disease activity (PtGDA) and physician global assessment of disease activity (PGDA) assessed on 0-10 centimeters (cm) visual analogue scale (VAS). Higher scores represent greater affectation due to disease activity. CDAI total score = 0-76. CDAI score less than or equal to (</=) 2.8 indicates disease remission, greater than (>) 2.8 to 10 indicates low disease activity, >10 to 22 indicates moderate disease activity, and >22 indicates high disease activity.
Time Frame: Baseline, Week 24
Population: FAS; Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 183
units on a scale | -21.6 (13.25)
Statistical Analysis 1: Comparison: Tocilizumab; Analysis for change from baseline to Week 24 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests

2. Primary Outcome: Change From Baseline in CDAI at Week 20
Description: The CDAI is a numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGDA and PGDA assessed on 0-10 cm VAS. Higher scores represent greater affectation due to disease activity. CDAI total score = 0-76. CDAI score </=2.8 indicates disease remission, >2.8 to 10 indicates low disease activity, >10 to 22 indicates moderate disease activity, and >22 indicates high disease activity.
Time Frame: Baseline, Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 185
units on a scale | -21.3 (12.87)

3. Primary Outcome: Change From Baseline in CDAI at Week 16
Description: as for outcome 2
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 191
units on a scale | -20.2 (12.53)

4. Primary Outcome: Change From Baseline in CDAI at Week 12
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 198
units on a scale | -19.1 (12.46)

5. Primary Outcome: Change From Baseline in CDAI at Week 8
Description: as for outcome 2
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 203
units on a scale | -17.7 (12.07)

6. Primary Outcome: Change From Baseline in CDAI at Week 4
Description: as for outcome 2
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 212
units on a scale | -14.0 (11.57)

7. Primary Outcome: Change From Baseline in CDAI at Week 2
Description: as for outcome 2
Time Frame: Baseline, Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 218
units on a scale | -9.1 (9.71)
Statistical Analysis 1: Comparison: Tocilizumab; Analysis for change from baseline to Week 2 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests

8. Secondary Outcome: Number of Participants Achieving Clinical Remission According to CDAI up to Week 52
Description: The CDAI is a numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGDA and PGDA assessed on 0-10 cm VAS. Higher scores represent greater affectation due to disease activity. CDAI total score = 0-76. CDAI score </=2.8 during any two consecutive visits, not including the baseline visit indicates disease remission.
Time Frame: Baseline up to Week 52 (Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 38, and 52)
Population: FAS
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 227
participants | 10

9. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count and Erythrocyte Sedimentation Rate (DAS28-ESR) at Weeks 2, 24, and 52
Description: DAS28-ESR is calculated from the TJC and SJC based on a 28-joint assessment, the erythrocyte sedimentation rate (ESR) in millimeters per hour (mm/hour) and PtGDA assessed on 0-10 cm VAS. Higher scores indicate greater affectation due to disease activity. DAS28-ESR total score= 0-9.4. DAS28-ESR </=3.2 indicates low disease activity, DAS28-ESR >3.2 to 5.1 indicates moderate to high disease activity, and DAS28-ESR </=3.2 indicates remission.
Time Frame: Baseline, Weeks 2, 24, and 52
Population: FAS; Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure and 'n' signifies the number of participants evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 216
units on a scale
  Baseline (n=216) | 5.81 (1.080)
  Change at Week 2 (n=208) | -1.5 (1.04)
  Change at Week 24 (n=174) | -3.2 (1.47)
  Change at Week 52 (n=31) | -3.6 (1.18)
Statistical Analysis 1: Comparison: Tocilizumab; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 2: Comparison: Tocilizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 3: Comparison: Tocilizumab; Analysis for change from baseline to Week 52 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests

10. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Weeks 2, 24, and 52
Description: SDAI is a numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PtGDA and PGDA assessed on 0-10 cm VAS and C-reactive protein (CRP) in milligrams per deciliter (mg/dL). Higher scores indicate greater affectation due to disease activity. SDAI total score = 0-86. SDAI </=3.3 indicates disease remission, >3.4 to 11 indicates low disease activity, >11 to 26 indicates moderate disease activity, and >26 indicates high disease activity.
Time Frame: Baseline, Weeks 2, 24, and 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 215
units on a scale
  Baseline (n=215) | 48.70 (45.790)
  Change at Week 2 (n=203) | -26.5 (44.04)
  Change at Week 24 (n=176) | -38.9 (48.75)
  Change at Week 52 (n=29) | -39.3 (26.82)
Statistical Analysis 1: Comparison: Tocilizumab; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 2: Comparison: Tocilizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 3: Comparison: Tocilizumab; [analysis description as in outcome 9, analysis 3]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests

11. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20), 50% (ACR50), and 70% (ACR70) Response
Description: The ACR 20, 50, and 70 responses: greater than or equal to (>/=) 20 percent (%), 50%, and 70% improvement in TJC and SJC (28 assessed joints), and 20%, 50%, 70% improvement in 3 of the following 5 criteria, respectively: 1) PGDA, 2) PtGDA, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) CRP or ESR at each visit.
Time Frame: Weeks 2, 24, and 52
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 222
percentage of participants
  Week 2: ACR 20 (n=222) | 18.5
  Week 2: ACR 50 (n=222) | 6.3
  Week 2: ACR 70 (n=222) | 11.7
  Week 24: ACR 20 (n=192) | 8.3
  Week 24: ACR 50 (n=192) | 4.7
  Week 24: ACR 70 (n=192) | 65.6
  Week 52: ACR 20 (n=70) | 0.0
  Week 52: ACR 50 (n=70) | 0.0
  Week 52: ACR 70 (n=70) | 40.0

12. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response Based on DAS28
Description: The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 </=3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to </=5.1 or change from baseline >0.6 to </=1.2 with DAS28 </=5.1; non-responders: change from baseline </=0.6 or change from baseline >0.6 and </=1.2 with DAS28 >5.1.
Time Frame: Baseline, Weeks 2, 24, and 52
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 222
percentage of participants
  Week 2: No Response (n=222) | 32.4
  Week 2: Moderate Response (n=222) | 50.5
  Week 2: Good Response (n=222) | 17.1
  Week 24: No Response (n=192) | 13.5
  Week 24: Moderate Response (n=192) | 25.0
  Week 24: Good Response (n=192) | 61.5
  Week 52: No Response (n=70) | 55.7
  Week 52: Moderate Response (n=70) | 8.6
  Week 52: Good Response (n=70) | 35.7

13. Secondary Outcome: Change From Baseline in Total TJC at Weeks 2, 24, and 52
Description: TJC was defined as the total number of painful joints based on 68-joint assessment (TJC-68) and 28-joint assessment (TJC-28).
Time Frame: Baseline, Weeks 2, 24, and 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 224
tender joints
  TJC-68, Baseline (n=223) | 16.91 (10.860)
  TJC-68, Change at Week 2 (n=218) | -5.4 (8.38)
  TJC-68, Change at Week 24 (n=188) | -12.9 (11.18)
  TJC-68, Change at Week 52 (n=69) | -16.5 (10.35)
  TJC-28, Baseline (n=224) | 11.32 (6.241)
  TJC-28, Change at Week 2 (n=219) | -3.7 (5.40)
  TJC-28, Change at Week 24 (n=189) | -8.6 (6.62)
  TJC-28, Change at Week 52 (n=70) | -11.0 (6.14)
Statistical Analysis 1: Comparison: Tocilizumab; TJC-68: Analysis for change from baseline to Week 2 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 2: Comparison: Tocilizumab; TJC-68: Analysis for change from baseline to Week 24 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 3: Comparison: Tocilizumab; TJC-68: Analysis for change from baseline to Week 52 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 4: Comparison: Tocilizumab; TJC-28: Analysis for change from baseline to Week 2 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 5: Comparison: Tocilizumab; TJC-28: Analysis for change from baseline to Week 24 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 6: Comparison: Tocilizumab; TJC-28: Analysis for change from baseline to Week 52 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests

14. Secondary Outcome: Change From Baseline in Total SJC at Weeks 2, 24, and 52
Description: SJC was defined as the total number of swollen joints based on 66-joint assessment (SJC-66) and 28-joint assessment (SJC-28).
Time Frame: Baseline, Weeks 2, 24, and 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 224
swollen joints
  SJC-66, Baseline (n=223) | 9.53 (6.713)
  SJC-66, Change at Week 2 (n=218) | -3.7 (4.94)
  SJC-66, Change at Week 24 (n=188) | -8.3 (6.73)
  SJC-66, Change at Week 52 (n=69) | -9.1 (6.66)
  SJC-28, Baseline (n=224) | 7.90 (5.203)
  SJC-28, Change at Week 2 (n=219) | -2.9 (3.91)
  SJC-28, Change at Week 24 (n=189) | -6.7 (5.17)
  SJC-28, Change at Week 52 (n=70) | -7.6 (4.63)
Statistical Analysis 1: Comparison: Tocilizumab; SJC-66: Analysis for change from baseline to Week 2 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 2: Comparison: Tocilizumab; SJC-66: Analysis for change from baseline to Week 24 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 3: Comparison: Tocilizumab; SJC-66: Analysis for change from baseline to Week 52 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 4: Comparison: Tocilizumab; SJC-28: Analysis for change from baseline to Week 2 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 5: Comparison: Tocilizumab; SJC-28: Analysis for change from baseline to Week 24 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 6: Comparison: Tocilizumab; SJC-28: Analysis for change from baseline to Week 52 was performed using Wilcoxon Rank Sum and Signed Rank Tests for dependent sample; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests

15. Secondary Outcome: Association Between Disease Activity Parameters: DAS28-ESR and CDAI, Assessed Using Correlation Coefficient
Description: DAS28-ESR is calculated from the TJC and SJC based on a 28-joint assessment, the ESR in mm/hour and PtGDA. DAS28-ESR total score= 0-9.4. Higher scores indicate greater affectation due to disease activity. The CDAI is a numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGDA and PGDA assessed on 0-10 cm VAS. CDAI total score = 0-76. Higher scores represent greater affectation due to disease activity. Correlation coefficient for relationship between DAS28-ESR and CDAI at different time points is reported. Correlation coefficient value range= -1 to 1. Higher positive value indicates greater positive relationship and higher negative value indicates greater negative relationship.
Time Frame: Weeks 2, 24, 52
Population: as for outcome 9
Measure: Number; unit: correlation coefficient
Arm/Group | Tocilizumab
Number analyzed (Participants) | 213
correlation coefficient
  Week 2 (n=213) | 0.86514
  Week 24 (n=182) | 0.86944
  Week 52 (n=32) | 0.87301
Statistical Analysis 1: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and CDAI at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and CDAI at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and CDAI at Week 52; Test type: Superiority or Other; p < 0.0001, ANOVA

16. Secondary Outcome: Association Between Disease Activity Parameters: DAS28-ESR and SDAI, Assessed Using Correlation Coefficient
Description: DAS28-ESR is calculated from the TJC and SJC based on a 28-joint assessment, the ESR in mm/hour and PtGDA. DAS28-ESR total score= 0-9.4. Higher scores indicate greater affectation due to disease activity. SDAI is a numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PtGDA and PGDA assessed on 0-10 cm VAS and CRP in mg/dL. SDAI total score= 0-86. Higher scores indicate greater affectation due to disease activity. Correlation coefficient for relationship between DAS28-ESR and SDAI at different time points is reported. Correlation coefficient value range= -1 to 1. Higher positive value indicates greater positive relationship and higher negative value indicates greater negative relationship.
Time Frame: Weeks 2, 24, 52
Population: as for outcome 9
Measure: Number; unit: correlation coefficient
Arm/Group | Tocilizumab
Number analyzed (Participants) | 213
correlation coefficient
  Week 2 (n=213) | 0.88118
  Week 24 (n=182) | 0.87060
  Week 52 (n=31) | 0.81995
Statistical Analysis 1: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and SDAI at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and SDAI at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and SDAI at Week 52; Test type: Superiority or Other; p < 0.0001, ANOVA

17. Secondary Outcome: Association Between Disease Activity Parameters: CDAI and SDAI, Assessed Using Correlation Coefficient
Description: The CDAI is a numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGDA and PGDA assessed on 0-10 cm VAS. CDAI total score = 0-76. Higher scores represent greater affectation due to disease activity. SDAI is a numerical sum of 5 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGDA and PGDA assessed on 0-10 cm VAS and CRP in mg/dL. SDAI total score= 0-86. Higher scores indicate greater affectation due to disease activity. Correlation coefficient for relationship between CDAI and SDAI at different time points is reported. Correlation coefficient value range= -1 to 1. Higher positive value indicates greater positive relationship and higher negative value indicates greater negative relationship.
Time Frame: Weeks 2, 24, 52
Population: as for outcome 9
Measure: Number; unit: correlation coefficient
Arm/Group | Tocilizumab
Number analyzed (Participants) | 213
correlation coefficient
  Week 2 (n=213) | 0.98602
  Week 24 (n=185) | 0.97515
  Week 52 (n=31) | 0.97389
Statistical Analysis 1: Comparison: Tocilizumab; Analysis for association between CDAI and SDAI at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab; Analysis for association between CDAI and SDAI at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab; Analysis for association between CDAI and SDAI at Week 52; Test type: Superiority or Other; p < 0.0001, ANOVA

18. Secondary Outcome: Association Between Disease Activity Parameter (DAS28-ESR) and Treatment Response Parameters (ACR20, ACR50, and ACR70), Assessed Using Regression Coefficient
Description: DAS28-ESR is calculated from the TJC and SJC based on a 28-joint assessment, the ESR in mm/hour and PtGDA. DAS28-ESR total score= 0-9.4. The ACR 20, 50, and 70 responses: >/=20%, 50%, and 70% improvement in TJC and SJC, and 20%, 50%, 70% improvement in 3 of the following 5 criteria, respectively: 1) PGDA, 2) PtGDA, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) CRP at each visit. Regression coefficients for relationship between DAS28-ESR and ACR responses (ACR20, ACR50, and ACR70) at different time points are reported. Regression coefficient value range= not defined (any negative or positive value is possible). Higher positive value indicates greater extent of positive relationship and higher negative value indicates greater extent of negative relationship.
Time Frame: Weeks 2, 24, 52
Population: as for outcome 9
Measure: Number; unit: regression coefficient
Arm/Group | Tocilizumab
Number analyzed (Participants) | 213
regression coefficient
  Week 2: DAS28-ESR and ACR20 (n=213) | -1.02676
  Week 2: DAS28-ESR and ACR50 (n=213) | -1.31737
  Week 2: DAS28-ESR and ACR70 (n=213) | -1.50400
  Week 24: DAS28-ESR and ACR20 (n=182) | -1.71191
  Week 24: DAS28-ESR and ACR50 (n=182) | -1.54281
  Week 24: DAS28-ESR and ACR70 (n=182) | -1.43977
  Week 52: DAS28-ESR and ACR20 (n=32) | -2.05036
  Week 52: DAS28-ESR and ACR50 (n=32) | -2.05036
  Week 52: DAS28-ESR and ACR70 (n=32) | -2.05036
Statistical Analysis 1: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and ACR20 at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and ACR50 at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and ACR70 at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 4: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and ACR20 at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 5: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and ACR50 at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and ACR70 at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 7: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and ACR20 at Week 52; Test type: Superiority or Other; p = 0.0004, ANOVA
Statistical Analysis 8: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and ACR50 at Week 52; Test type: Superiority or Other; p = 0.0004, ANOVA
Statistical Analysis 9: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and ACR70 at Week 52; Test type: Superiority or Other; p = 0.0004, ANOVA

19. Secondary Outcome: Association Between Disease Activity Parameter (DAS28-ESR) and Treatment Response Parameter (EULAR), Assessed Using Regression Coefficient
Description: DAS28-ESR is calculated from the TJC and SJC based on a 28-joint assessment, the ESR in mm/hour and PtGDA. DAS28-ESR total score= 0-9.4. EULAR response criteria (based on DAS28 score): Good responders (change from baseline >1.2 with DAS28 </=3.2); Moderate responders (change from baseline >1.2 with DAS28 >3.2 to </=5.1 or change from baseline >0.6 to </=1.2 with DAS28 </=5.1); Non-responders (change from baseline </=0.6 or change from baseline >0.6 and </=1.2 with DAS28 >5.1). Regression coefficient for relationship between DAS28-ESR and EULAR Good response at different time points is reported. Regression coefficient value range= not defined (any negative or positive value is possible). Higher positive value indicates greater extent of positive relationship and higher negative value indicates greater extent of negative relationship.
Time Frame: Weeks 2, 24, 52
Population: as for outcome 9
Measure: Number; unit: regression coefficient
Arm/Group | Tocilizumab
Number analyzed (Participants) | 213
regression coefficient
  Week 2: DAS28-ESR and EULAR (n=213) | -1.62883
  Week 24: DAS28-ESR and EULAR (n=182) | -1.36226
  Week 52: DAS28-ESR and EULAR (n=32) | -1.47781
Statistical Analysis 1: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and EULAR at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and EULAR at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab; Analysis for association between DAS28-ESR and EULAR at Week 52; Test type: Superiority or Other; p < 0.0001, ANOVA

20. Secondary Outcome: Association Between Disease Activity Parameter (CDAI) and Treatment Response Parameters (ACR20, ACR50, and ACR70), Assessed Using Regression Coefficient
Description: The CDAI is a numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGDA and PGDA assessed on 0-10 cm VAS. CDAI total score = 0-76. The ACR 20, 50, and 70 responses: >/=20%, 50%, and 70% improvement in TJC and SJC, and 20%, 50%, 70% improvement in 3 of the following 5 criteria, respectively: 1) PGDA, 2) PtGDA, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) CRP at each visit. Regression coefficients for relationship between CDAI and ACR responses (ACR20, ACR50, and ACR70) at different time points are reported. Regression coefficient value range= not defined (any negative or positive value is possible). Higher positive value indicates greater extent of positive relationship and higher negative value indicates greater extent of negative relationship.
Time Frame: Weeks 2, 24, 52
Population: as for outcome 9
Measure: Number; unit: regression coefficient
Arm/Group | Tocilizumab
Number analyzed (Participants) | 220
regression coefficient
  Week 2: CDAI and ACR20 (n=220) | -9.65473
  Week 2: CDAI and ACR50 (n=220) | -10.67389
  Week 2: CDAI and ACR70 (n=220) | -13.38810
  Week 24: CDAI and ACR20 (n=186) | -13.18433
  Week 24: CDAI and ACR50 (n=186) | -11.95933
  Week 24: CDAI and ACR70 (n=186) | -11.18299
  Week 52: CDAI and ACR20 (n=32) | -18.94643
  Week 52: CDAI and ACR50 (n=32) | -18.94643
  Week 52: CDAI and ACR70 (n=32) | -18.94643
Statistical Analysis 1: Comparison: Tocilizumab; Analysis for association between CDAI and ACR20 at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab; Analysis for association between CDAI and ACR50 at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab; Analysis for association between CDAI and ACR70 at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 4: Comparison: Tocilizumab; Analysis for association between CDAI and ACR20 at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 5: Comparison: Tocilizumab; Analysis for association between CDAI and ACR50 at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: Tocilizumab; Analysis for association between CDAI and ACR70 at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 7: Comparison: Tocilizumab; Analysis for association between CDAI and ACR20 at Week 52; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 8: Comparison: Tocilizumab; Analysis for association between CDAI and ACR50 at Week 52; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 9: Comparison: Tocilizumab; Analysis for association between CDAI and ACR70 at Week 52; Test type: Superiority or Other; p < 0.0001, ANOVA

21. Secondary Outcome: Association Between Disease Activity Parameter (CDAI) and Treatment Response Parameter (EULAR), Assessed Using Regression Coefficient
Description: The CDAI is a numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGDA and PGDA assessed on 0-10 cm VAS. CDAI total score = 0-76. EULAR response criteria (based on DAS28 score): Good responders (change from baseline >1.2 with DAS28 </=3.2); Moderate responders (change from baseline >1.2 with DAS28 >3.2 to </=5.1 or change from baseline >0.6 to </=1.2 with DAS28 </=5.1); Non-responders (change from baseline </=0.6 or change from baseline >0.6 and </=1.2 with DAS28 >5.1). Regression coefficient for relationship between CDAI and EULAR Good response at different time points is reported. Regression coefficient value range= not defined (any negative or positive value is possible). Higher positive value indicates greater extent of positive relationship and higher negative value indicates greater extent of negative relationship.
Time Frame: Weeks 2, 24, 52
Population: as for outcome 9
Measure: Number; unit: regression coefficient
Arm/Group | Tocilizumab
Number analyzed (Participants) | 220
regression coefficient
  Week 2: CDAI and EULAR (n=220) | -10.97686
  Week 24: CDAI and EULAR (n=186) | -7.03184
  Week 52: CDAI and EULAR (n=32) | -9.46563
Statistical Analysis 1: Comparison: Tocilizumab; Analysis for association between CDAI and EULAR at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab; Analysis for association between CDAI and EULAR at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab; Analysis for association between CDAI and EULAR at Week 52; Test type: Superiority or Other; p < 0.0001, ANOVA

22. Secondary Outcome: Association Between Disease Activity Parameter (SDAI) and Treatment Response Parameters (ACR20, ACR50, and ACR70), Assessed Using Regression Coefficient
Description: SDAI is a numerical sum of 5 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGDA and PGDA assessed on 0-10 cm VAS and CRP in mg/dL. SDAI total score= 0-86. The ACR 20, 50, and 70 responses: >/=20%, 50%, and 70% improvement in TJC and SJC, and 20%, 50%, 70% improvement in 3 of the following 5 criteria, respectively: 1) PGDA, 2) PtGDA, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) CRP at each visit. Regression coefficients for relationship between SDAI and ACR responses (ACR20, ACR50, and ACR70) at different time points are reported. Regression coefficient value range= not defined (any negative or positive value is possible). Higher positive value indicates greater extent of positive relationship and higher negative value indicates greater extent of negative relationship.
Time Frame: Weeks 2, 24, 52
Population: as for outcome 9
Measure: Number; unit: regression coefficient
Arm/Group | Tocilizumab
Number analyzed (Participants) | 213
regression coefficient
  Week 2: SDAI and ACR20 (n=213) | -9.44923
  Week 2: SDAI and ACR50 (n=213) | -10.74230
  Week 2: SDAI and ACR70 (n=213) | -13.31421
  Week 24: SDAI and ACR20 (n=185) | -14.19790
  Week 24: SDAI and ACR50 (n=185) | -12.65454
  Week 24: SDAI and ACR70 (n=185) | -11.78067
  Week 52: SDAI and ACR20 (n=31) | -22.83519
  Week 52: SDAI and ACR50 (n=31) | -22.83519
  Week 52: SDAI and ACR70 (n=31) | -22.83519
Statistical Analysis 1: Comparison: Tocilizumab; Analysis for association between SDAI and ACR20 at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab; Analysis for association between SDAI and ACR50 at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab; Analysis for association between SDAI and ACR70 at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 4: Comparison: Tocilizumab; Analysis for association between SDAI and ACR20 at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 5: Comparison: Tocilizumab; Analysis for association between SDAI and ACR50 at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: Tocilizumab; Analysis for association between SDAI and ACR70 at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 7: Comparison: Tocilizumab; Analysis for association between SDAI and ACR20 at Week 52; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 8: Comparison: Tocilizumab; Analysis for association between SDAI and ACR50 at Week 52; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 9: Comparison: Tocilizumab; Analysis for association between SDAI and ACR70 at Week 52; Test type: Superiority or Other; p < 0.0001, ANOVA

23. Secondary Outcome: Association Between Disease Activity Parameter (SDAI) and Treatment Response Parameter (EULAR), Assessed Using Regression Coefficient
Description: The SDAI is a numerical sum of 5 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGDA and PGDA assessed on 0-10 cm VAS and CRP in mg/dL. SDAI total score= 0-86. EULAR response criteria (based on DAS28 score): Good responders (change from baseline >1.2 with DAS28 </=3.2); Moderate responders (change from baseline >1.2 with DAS28 >3.2 to </=5.1 or change from baseline >0.6 to </=1.2 with DAS28 </=5.1); Non-responders (change from baseline </=0.6 or change from baseline >0.6 and </=1.2 with DAS28 >5.1). Regression coefficient for relationship between SDAI and EULAR Good response at different time points is reported. Regression coefficient value range= not defined (any negative or positive value is possible). Higher positive value indicates greater extent of positive relationship and higher negative value indicates greater extent of negative relationship.
Time Frame: Weeks 2, 24, 52
Population: as for outcome 9
Measure: Number; unit: regression coefficient
Arm/Group | Tocilizumab
Number analyzed (Participants) | 213
regression coefficient
  Week 2: SDAI and EULAR (n=213) | -11.73463
  Week 24: SDAI and EULAR (n=185) | -7.32435
  Week 52: SDAI and EULAR (n=31) | -9.64146
Statistical Analysis 1: Comparison: Tocilizumab; Analysis for association between SDAI and EULAR at Week 2; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab; Analysis for association between SDAI and EULAR at Week 24; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab; Analysis for association between SDAI and EULAR at Week 52; Test type: Superiority or Other; p = 0.0016, ANOVA

24. Secondary Outcome: Percentage of DMARDs Dose Reductions and/or Discontinuation Events by Reasons
Description: Percentage of DMARDs dose reduction and/or discontinuation (Red/Dis) events is reported by different reasons.
Time Frame: Baseline up to Week 52
Population: FAS; Here, 'Overall Number of Participants Analyzed' signifies the number of participants with DMARDs dose reductions and/or discontinuation.
Measure: Number; unit: percentage of events
Units Other Than Participants: DMARDs Dose Red/Dis Events
Arm/Group | Tocilizumab
Number analyzed (Participants) | 79
Number analyzed (DMARDs Dose Red/Dis Events) | 148
percentage of events
  Safety | 27.7
  Discomfort | 9.5
  Lack of Efficacy | 29.7
  Other Than Above | 31.1
  Unknown | 2.0

25. Secondary Outcome: Percentage of Non-DMARDs Dose Reductions and/or Discontinuation Events by Reasons
Description: Percentage of Non-DMARDs dose reduction and/or discontinuation (Red/Dis) events is reported by different reasons.
Time Frame: Baseline up to Week 52
Population: FAS; Here, 'Overall Number of Participants Analyzed' signifies the number of participants with non-DMARDs dose reductions and/or discontinuation.
Measure: Number; unit: percentage of events
Units Other Than Participants: Non-DMARDs Dose Red/Dis Events
Arm/Group | Tocilizumab
Number analyzed (Participants) | 154
Number analyzed (Non-DMARDs Dose Red/Dis Events) | 547
percentage of events
  Safety | 9.5
  Discomfort | 1.3
  Lack of Efficacy | 8.8
  Other Than Above | 73.7
  Unknown | 6.8

26. Secondary Outcome: Change From Baseline in PtGDA VAS Score at Weeks 2, 24, and 52
Description: Participants answered the following question: "Considering all the ways your arthritis affects you, how are you feeling today." Participants responded by using a 0 - 100 millimeter (mm) VAS, where 0 mm = very well and 100 mm = very poorly.
Time Frame: Baseline, Weeks 2, 24, and 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 226
mm
  Baseline (n=226) | 61.31 (23.526)
  Change at Week 2 (n=220) | -10.6 (20.99)
  Change at Week 24 (n=186) | -28.4 (27.40)
  Change at Week 52 (n=32) | -38.4 (27.65)
Statistical Analysis 1: Comparison: Tocilizumab; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 2: Comparison: Tocilizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 3: Comparison: Tocilizumab; [analysis description as in outcome 9, analysis 3]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests

27. Secondary Outcome: Change From Baseline in PGDA VAS Score at Weeks 2, 24, and 52
Description: The physician assessed participant's current disease activity on a 0-100 mm VAS, where 0 mm = no disease activity and 100 mm = maximum disease activity.
Time Frame: Baseline, Weeks 2, 24, and 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 226
mm
  Baseline (n=226) | 57.36 (19.228)
  Change at Week 2 (n=220) | -15.3 (17.49)
  Change at Week 24 (n=186) | -38.0 (25.13)
  Change at Week 52 (n=32) | -43.9 (17.13)
Statistical Analysis 1: Comparison: Tocilizumab; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 2: Comparison: Tocilizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 3: Comparison: Tocilizumab; [analysis description as in outcome 9, analysis 3]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests

28. Secondary Outcome: Participant Pain VAS Score at Weeks 2, 24, and 52
Description: Participants assessed their pain using a 0-100 mm VAS. Intensity of pain range (over past week): 0 mm = no pain to 100 mm = worst possible pain.
Time Frame: Weeks 2, 24, and 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 226
mm
  Baseline (n=226) | 58.21 (23.622)
  Change at Week 2 (n=220) | -11.4 (22.38)
  Change at Week 24 (n=186) | -26.5 (27.31)
  Change at Week 52 (n=32) | -36.0 (26.82)
Statistical Analysis 1: Comparison: Tocilizumab; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 2: Comparison: Tocilizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 3: Comparison: Tocilizumab; [analysis description as in outcome 9, analysis 3]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests

29. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Weeks 2, 24, and 52
Description: HAQ-DI is a participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Weeks 2, 24, and 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 223
units on a scale
  Baseline (n=223) | 1.04 (0.687)
  Change at Week 2 (n=215) | -0.2 (0.44)
  Change at Week 24 (n=183) | -0.4 (0.63)
  Change at Week 52 (n=31) | -0.5 (0.69)
Statistical Analysis 1: Comparison: Tocilizumab; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 2: Comparison: Tocilizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 3: Comparison: Tocilizumab; [analysis description as in outcome 9, analysis 3]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests

30. Secondary Outcome: Missed Working Days Assessed Using Short Form-Health and Labor Questionnaire (SF-HLQ) Score at Weeks 24 and 52
Description: The SF-HLQ assessed productivity losses related to health problems in individuals with paid or unpaid work and consisted of three modules (absenteeism from paid work, production losses without absenteeism from paid work and hindrance in the performance of paid and unpaid work). Any missed working days or number of worked days with reduced efficiency during the last month were reported.
Time Frame: Weeks 24 and 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tocilizumab
Number analyzed (Participants) | 69
days
  Week 24 (n=69) | 6.4 (45.09)
  Week 52 (n=7) | 0.3 (0.76)

31. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) Total Score at Weeks 2, 24, and 52
Description: FACIT total score is sum of Functional Assessment of Cancer Therapy-General (FACT-G) score and Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F; additional concerns) score. FACT-G is a core questionnaire that evaluates quality of life (QoL) in cancer population. FACT-G consists of 27 questions grouped in 4 domains of general health-related QoL: physical well-being, social/family well-being, emotional well-being, and functional well-being; each item ranges from 0 (not at all) to 4 (very much). FACT-G score ranges between 0-108. FACIT-F is a 13-item questionnaire that evaluates self-reported fatigue and its impact upon daily activities. Each item ranges from 0 (Not at all) to 4 (Very much). The sum of all responses result in the FACIT total score with a total possible range of 0 (better score) to 160 (worse score). Negative change from baseline represents a better QoL.
Time Frame: Baseline, Weeks 2, 24, and 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 207
units on a scale
  Baseline (n=207) | 72.41 (16.806)
  Change at Week 2 (n=196) | -5.8 (14.10)
  Change at Week 24 (n=165) | -11.1 (18.60)
  Change at Week 52 (n=60) | -43.8 (34.87)
Statistical Analysis 1: Comparison: Tocilizumab; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 2: Comparison: Tocilizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 3: Comparison: Tocilizumab; [analysis description as in outcome 9, analysis 3]; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum and Signed Rank Tests

32. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) at Weeks 24 and 52
Description: PSQI is a questionnaire with 18 questions to assess sleep quality. The 18 questions are distributed to 7 elements (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction). A participant indicates how frequently each item was experienced on a scale from 0 to 3. The global score is the sum score of all 7 elements and ranges from 0-21 with higher values indicating worse sleep quality. A score of >/=5 indicates poor sleepers.
Time Frame: Baseline, Weeks 24 and 52
Population: Per-protocol analysis set (PPAS) included all participants in FAS without any major protocol violation and who completed 24 weeks of treatment period. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome; 'n'=participants evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 103
units on a scale
  Baseline (n=103) | 11.00 (2.719)
  Change at Week 24 (n=73) | -0.7 (2.39)
  Change at Week 52 (n=16) | -0.9 (2.42)
Statistical Analysis 1: Comparison: Tocilizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0045, Wilcoxon Rank Sum and Signed Rank Tests
Statistical Analysis 2: Comparison: Tocilizumab; [analysis description as in outcome 9, analysis 3]; Test type: Superiority or Other; p = 0.1992, Wilcoxon Rank Sum and Signed Rank Tests

33. Secondary Outcome: Treatment Compliance, as Assessed Using Participant Diary Cards and Return Records
Description: Treatment Compliance was calculated as (total actual doses taken for the period) / (total planned or prescribed dose for the period) x 100.
Time Frame: Weeks 24 and 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of planned dose
Arm/Group | Tocilizumab
Number analyzed (Participants) | 222
percentage of planned dose
  Week 24 (n=221) | 94.9 (10.20)
  Week 52 (n=222) | 94.7 (10.12)

34. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) of Special Interest
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs are AEs occurring between the first dose of study drug and up to 28 days after the last dose that were absent before treatment or that worsened relative to pre-treatment state. Following AEs were considered as AEs of special interest: anaphylactic reaction, hypersensitivity, stress cardiomyopathy, Gilbert's syndrome, gastrointestinal perforation, injection site erythema, injection site hypersensitivity, injection site irritation, injection site pruritus, arthritis bacterial, cellulitis, klebsiella infection, oral candidiasis, pneumonia, skin infection, vulvovaginal candidiasis, alanine aminotransferase increased, hepatic enzyme increased, brain neoplasm malignant, and urticaria.
Time Frame: Baseline up to 95 weeks
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 227
percentage of participants | 7.5

35. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATA) to Tocilizumab
Description: Percentage of participants with positive results for ATA against tocilizumab at different time points is reported.
Time Frame: Baseline, Weeks 12, 24, 38, 52, at 8 weeks after last dose (up to Week 60), at early withdrawal (up to Week 52), at Follow-up Visits 1 (Week 64), 2 (Week 76), and 3 (Week 88)
Population: FAS; Here, 'n' signifies the number of participants evaluable at specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 227
percentage of participants
  Baseline (n=227) | 2.6
  Week 12 (n=6) | 100.0
  Week 24 (n=179) | 1.7
  Week 38 (n=6) | 33.3
  Week 52 (n=161) | 1.2
  8 Weeks After Last Dose (up to Week 60) (n=41) | 2.4
  Early Withdrawal (up to Week 52) (n=31) | 6.5
  Follow-up Visit 1 (Week 64) (n=16) | 100.0
  Follow-up Visit 2 (Week 76) (n=11) | 100.0
  Follow-up Visit 3 (Week 88) (n=3) | 100.0

36. Secondary Outcome: Mean Tocilizumab Concentration
Time Frame: Baseline, Weeks 12, 24, 38, 52, at early withdrawal (up to Week 52), at Follow-up Visit 2 (Week 76)
Population: FAS; Here 'n' signifies the number of participants evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 227
micrograms per milliliter (mcg/mL)
  Baseline (n=2) | 35.6 (48.89)
  Week 12 (n=186) | 46.4 (23.01)
  Week 24 (n=177) | 52.6 (28.21)
  Week 38 (n=169) | 55.2 (30.55)
  Week 52 (n=165) | 54.0 (29.00)
  Early Withdrawal (up to Week 52) (n=19) | 24.8 (22.90)
  Follow-up Visit 2 (Week 76) (n=17) | 49.2 (34.05)

37. Secondary Outcome: Mean Soluble Interleukin-6 Receptor (sIL-6R) Concentration
Time Frame: Baseline, Weeks 12, 24, 38, 52, at early withdrawal (up to Week 52), at Follow-up Visit 2 (Week 76)
Population: FAS; Here 'n' signifies the number of participants evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 227
nanograms per milliliter (ng/mL)
  Baseline (n=213) | 43.6 (49.30)
  Week 12 (n=189) | 543.9 (144.34)
  Week 24 (n=181) | 536.3 (144.32)
  Week 38 (n=171) | 557.8 (144.23)
  Week 52 (n=168) | 539.4 (147.04)
  Early Withdrawal (up to Week 52) (n=32) | 329.1 (257.30)
  Follow-up Visit 2 (Week 76) (n=18) | 523.4 (161.14)

ADVERSE EVENTS:
Time Frame: Day 1 up to approximately 95 weeks
Description: FAS; TEAEs are adverse events occurring between the first dose of study drug and up to 28 days after the last dose that were absent before treatment or that worsened relative to pre-treatment state.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 17/227
Other Adverse Events (participants affected / at risk) | 36/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=227)
Stress cardiomyopathy (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Carcinoembryonic antigen increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Aneurysm (Vascular disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Device breakage (Product Issues) | 1
Bladder neoplasm surgery (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=227)
Influenza (Infections and infestations) | 23
Transaminases increased (Investigations) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Bronchitis (Infections and infestations) | 15
Urinary tract infection (Infections and infestations) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.